CLINICAL TRIAL: NCT02856828
Title: Novel Use of an Enhanced Fluoroscopic Imaging Device to Reduce Radiation Exposure and Operative Time During Intramedullary Nailing of Hip Fractures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Closed due to slow enrollment.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00074745
Record Dates: First submitted 2016-07-28; First posted 2016-08-05 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Radiation Exposure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Digital Image Enhancement (DIE) Group (Experimental): A novel digital image enhancement technology will be used intraoperatively
  Interventions: Device: DIE
- Control Group (No Intervention): Standard intraoperative imaging will be used intraoperatively

INTERVENTIONS:
Device: DIE — digital image enhancement
  Arms: Digital Image Enhancement (DIE) Group

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a novel digital image enhancement (DIE) technology in reducing the radiation exposure to both the patient and surgical staff during standard intramedullary nail placement for treatment of hip fractures. Secondarily, to evaluate whether the image quality and reproducibility of desired images can be improved with use of the DIE technology. Finally, to evaluate whether DIE technology reduces total operative time.

ELIGIBILITY:
Inclusion Criteria:

* closed hip fracture requiring intramedullary nailing

Exclusion Criteria:

* age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-02-06 (Actual); Study Completion 2018-02-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Digital Image Enhancement (DIE) Group | Control Group
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Hip fracture patients only, not surgeons
Groups:
- Total: Total of all reporting groups
Arm/Group | Digital Image Enhancement (DIE) Group | Control Group | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 0 | 1 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Radiation Exposure to Patient During Intramedullary Nail Placement for Treatment of Hip Fractures as Measured by Dosimeter Badge
Time Frame: intraoperatively
Measure: Number; unit: mGy
Groups:
- Digital Image Enhancement (DIE) Group: The radiation exposure to the patient in the digital image enhancement group.
- Control Group: The radiation exposure to the patient in the standard intraoperative imaging group.
Arm/Group | Digital Image Enhancement (DIE) Group | Control Group
Number analyzed (Participants) | 2 | 3
mGy
  Participant 1 | 5.12 | NA — Participant was in the DIE Group.
  Participant 2 | NA — Participant was in the Control Group. | 12.9
  Participant 3 | 9.79 | NA — Participant was in the DIE Group.
  Participant 4 | NA — Participant was in the Control Group. | 7.93
  Participant 5 | NA — Participant was in the Control Group. | 15.41

2. Primary Outcome: Radiation Exposure to Surgeon During Intramedullary Nail Placement for Treatment of Hip Fractures as Measured by Dosimeter Badge
Time Frame: intraoperatively
Measure: Number; unit: mrem
Groups:
- Digital Image Enhancement (DIE) Group: The radiation exposure to the primary surgeon of the participants from the novel digital image enhancement group.
- Control Group: The radiation exposure of the primary surgeon of the participants in the standard intraoperative imaging group.
Arm/Group | Digital Image Enhancement (DIE) Group | Control Group
Number analyzed (Participants) | 2 | 3
mrem
  Primary Surgeon 1 | 0.7 | NA — This participant was not in the control group.
  Primary Surgeon 2 | NA — This participant was not in the Digital Image Enhancement group. | 1.9
  Primary Surgeon 3 | 1.6 | NA — This participant was not in the control group.
  Primary Surgeon 4 | NA — This participant was not in the Digital Image Enhancement group. | 1.2
  Primary Surgeon 5 | NA — This participant was not in the Digital Image Enhancement group. | 3.1

3. Primary Outcome: Radiation Exposure to Scrub Tech During Intramedullary Nail Placement for Treatment of Hip Fractures as Measured by Dosimeter Badge
Time Frame: intraoperatively
Measure: Number; unit: mrem
Groups:
- Digital Image Enhancement (DIE) Group: The radiation exposure to the surgical technician of the participants from the novel digital image enhancement group.
- Control Group: The radiation exposure of the surgical technician of the participants in the standard intraoperative imaging group.
Arm/Group | Digital Image Enhancement (DIE) Group | Control Group
Number analyzed (Participants) | 2 | 3
mrem
  Surgical Technician 1 | 0.5 | NA — This participant was not in the Control group.
  Surgical Technician 2 | NA — This participant was not in the Digital Image Enhancement group. | 1.1
  Surgical Technician 3 | 0.9 | NA — This participant was not in the Control group.
  Surgical Technician 4 | NA — This participant was not in the Digital Image Enhancement group. | 0.9
  Surgical Technician 5 | NA — This participant was not in the Digital Image Enhancement group. | 0.1

4. Secondary Outcome: Image Quality and Reproducibility of Desired Images
Description: Measured by questionnaire related to image quality. Quality scale of 1-10, 1 being poor image quality and 10 being excellent image quality.
Time Frame: intraoperatively
Measure: Number; unit: Quality Scale of 1-10, 10 being the best
Groups:
- Image Quality of the Digital Image Enhancement (DIE) Group: The image quality, on a scale of 1-10 with 10 being the best quality, obtained for the novel digital image enhancement technology that was used intraoperatively.
  DIE: digital image enhancement
- Image Quality of the Control Group: The image quality, on a scale of 1-10 with 10 being the best quality, obtained for the standard intraoperative imaging that was used intraoperatively.
Arm/Group | Image Quality of the Digital Image Enhancement (DIE) Group | Image Quality of the Control Group
Number analyzed (Participants) | 2 | 3
Quality Scale of 1-10, 10 being the best
  Participant 1 Image | 9 | NA — This participant was not in the Control group.
  Participant 2 Image | NA — This participant was not in the Digital Image Enhancement group. | 8
  Participant 3 Image | 8 | NA — This participant was not in the Control group.
  Participant 4 Image | NA — This participant was not in the Digital Image Enhancement group. | 7
  Participant 5 Image | NA — This participant was not in the Digital Image Enhancement group. | 9

5. Secondary Outcome: Operative Time
Time Frame: intraoperatively
Measure: Number; unit: minutes
Groups:
- Digital Image Enhancement (DIE) Group: Operative time of the participants in the Digital Image Enhancement Group.
- Control Group: Operative time of the participants in the Standard Intraoperative Group.
Arm/Group | Digital Image Enhancement (DIE) Group | Control Group
Number analyzed (Participants) | 2 | 3
minutes
  Participant 1 | 51 | NA — This participant was not in the Control group.
  Participant 2 | NA — This participant was not in the Digital Image Enhancement group. | 103
  Participant 3 | 79 | NA — This participant was not in the Control group.
  Participant 4 | NA — This participant was not in the Digital Image Enhancement group. | 80
  Participant 5 | NA — This participant was not in the Digital Image Enhancement group. | 125

ADVERSE EVENTS:
Time Frame: During surgery and post-operative time of hospital admission, approximately 2 days
Arm/Group | Digital Image Enhancement (DIE) Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 0/2 | 0/3

LIMITATIONS AND CAVEATS:
Only two radiation dosimeters were purchased. Therefore, there is no radiation exposure data for the secondary surgeon.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-29): https://cdn.clinicaltrials.gov/large-docs/28/NCT02856828/Prot_SAP_000.pdf